CLINICAL TRIAL: NCT07155993
Title: FastForward: A Prospective Analysis of Long-term Fasting and Subsequent Food Reintroduction in Humans
Acronym: FastForward
Status: Enrolling by invitation | Type: Observational
Sponsor: Buchinger Wilhelmi Development & Holding GmbH (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Principal Investigator, Andrea Siegler, MD, Principal Investigator, Buchinger Wilhelmi Development & Holding GmbH
Other Study IDs: F-2024-032
Record Dates: First submitted 2025-07-23; First posted 2025-09-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetes (DM); Pre Diabetes; Overweight (BMI > 25)
Keywords: long-term fasting; fasting; continuous glucose monitoring; food reintroduction; meal documentation
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Overweight; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples With DNA — This study involves the collection and retention of the following biospecimens:
  Venous whole blood (liquid samples): Collected via standard venipuncture into during fasting and follow-up timepoints to assess metabolic, hormonal, and inflammatory biomarkers.
  Capillary blood (dried blood spot samples): Self-collected by participants in the clinic and at home using finger-prick methods and spotted onto a collection fdevice. These samples are used for remote monitoring of selected biomarkers including HbA1c.
  Stool samples: Self-collected by participants in the clinic and at home using standardized kits.
  All biospecimens are retained for future analysis of physiological responses to long-term fasting and the food reintroduction phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Food reintroduction observation group: Participants undergo a supervised long-term fast (≥5 days) followed by a structured food reintroduction at the Buchinger Wilhelmi Clinic. All participants complete online questionnaires assessing dietary habits, weight, and well-being during fasting and for up to 3 months afterward. Participants are monitored closely during the initial 14 days post-fasting with continuous glucose monitoring (CGM), photo-based meal tracking, and at-home dried blood spot sampling. Liquid venous blood and stool samples are collected at defined timepoints to analyze metabolic and physiological responses to fasting and food reintroduction.

SUMMARY:
This study explores what happens in the body and wellbeing during and after a period of long-term fasting. At the Buchinger Wilhelmi Clinic, participants follow a medically supervised fasting program lasting five or more days, followed by a structured food reintroduction phase. The study observes participants over time to better understand how fasting and the return to eating affect weight, metabolism, nutrition habits, and overall well-being.

All participants will complete online questionnaires during the fasting phase and for up to three months afterward. These surveys help track changes in lifestyle, mood, and health. In addition during the first two weeks after fasting ends participants wear a continuous glucose monitor (CGM) to track blood sugar levels in real time, use a mobile app to document meals with photos, and perform simple at-home blood tests using dried blood spot (DBS) kits.

By combining digital tools with personal reports and at home tests, the study aims to gain a clearer picture of how the body adapts after a prolonged fast. The goal is to better understand the short- and medium-term effects of extended fasting on metabolism, diet, and well-being-and to provide practical guidance for those interested in fasting as a health practice.

DETAILED DESCRIPTION:
Dear prospective study participants,

For optimal results of a fasting cure, the investigators would like to better understand the phase of food reintroduction, in which food is taken back after fasting.

The investigators would like to ask potential participants if they are willing to participate in the study of the Buchinger Wilhelmi Fasting Program. The study examines the post-fasting phase of food reintroduction. For this purpose, the first 14 days after the end of the fast are closely documented. This is done with the help of continuous glucose measurement and documentation of meals. In addition, various systemic biomarkers and the inflammatory status in blood are examined. In addition, further follow-up examinations take place after one and three months.

This study will include a total of more than 200 participants.

How will the study proceed and what investigations are planned?

The stay in the clinic begins with the admission examination by the study doctor, who explains the course of the study in detail and asks participants to sign the consent form. On the day of arrival, participants will receive an organic vegetarian dinner. This is followed by a "digestive rest day", a transitional day that is intended to prepare the body for the fasting phase. It consists of an easily digestible low-calorie mono-diet in three portions.

The fasting phase begins with a colon cleanse, e.g. with Glauber's salt. During fasting, the daily food intake consists of 1/4 l of freshly squeezed fruit or vegetable juice or 1/4 l of vegetable broth at noon, 1/4 l of vegetable broth in the evening and optionally 20 g of honey throughout the day. The end of fasting occurs individually after 7 or more (7+) days and is complemented by a phase of slow reintroduction of food with an ovo-lacto-vegetarian diet.

The study participants are offered the usual program of the Buchinger Wilhelmi Clinic. This includes fasting, physical exercise and individual treatments.

In addition to the admission examination, examinations take place during the clinic stay at the end of the fast and at the end of the food reintroduction.

The follow-up examinations 7, 14 and 21 days, one and three months after fasting take place independently from home. For study participants who live in the vicinity of the Buchinger Wilhelmi Clinic, the follow-up examinations take place after 14 days, one and three months on site at the Buchinger Wilhelmi Clinic in order to collect anthropometric data and take venous blood samples. If this applies to a participant, they will be contacted by the investigators.

If participants return to the clinic within 3 to 18 months after their initial stay, the investigators would carry out a follow-up examination including anthropometric measurements and a venous blood draw.

The following examinations will be carried out as part of the study:

Filling out questionnaires:

Participants will be asked about their lifestyle, their general health and their mental well-being before and at the end of the fast, at the end of the food reintroduction, 7, 14 and 21 days as well as one and three months after the fast. This will take about 15 minutes. During the fasting days and the first 14 days after fasting, participants will be asked daily about their well-being (approx. 5 minutes). All questionnaires are provided via the Buchinger Wilhelmi Amplius app and filled out in the app.

Documentation of anthropometric data:

During the stay, body weight, blood pressure and heart rate are measured daily in the morning by the nursing staff. The data is also recorded 7, 14 and 21 days, as well as one and three months after fasting through self-documentation. For this purpose, the body weight is measured at home on the scales. Blood pressure and heart rate are only measured at home if the appropriate devices are available. All values measured at home are entered into the Buchinger Wilhelmi Amplius app (there are fields in the questionnaires for this).

The waist circumference is measured at the beginning and end of fasting.

A bioelectrical impedance analysis (BIA) measurement takes place before fasting in the clinic. If participants come to the clinic for follow-up examinations, the measurement will take place again 14 days, one and three months after fasting. In BIA, body composition is measured by means of a weak current flow, which determines the percentage of muscle and fat mass in the body. The measurement must not be carried out in people with a pacemaker (tell the study doctor if this applies).

Blood analysis:

During the study, at least three, up to six, venous blood samples will be taken. On the first morning of the stay and at the end of the 7+ fasting days, as well as 3±2 days after breaking the fast, up to 30 ml of blood (amount of 2 tablespoons) is taken.

In addition, a total of 4 capillary blood samples are collected. On the first morning of the stay, as well as 14 days, one and three months after fasting. A small amount of blood is collected on blood collection swabs by a small prick in the fingertip. The capillary blood samples at the times after fasting must be taken by the participant themrselves with the equipment provided and sent by post to the research department of Buchinger Wilhelmi.

Blood sampling is a minimally invasive procedure in which a risk of side effects such as hematomas, infections, thrombosis or nerve damage cannot be ruled out.

Nutrition protocol:

From the day of breaking the fast, participants will log their meals for 14 days. To simplify this, the smartphone app "MyFoodRepo" is being used, developed by scientists for logging meals. This complies with the data protection guidelines of the GDPR. In the app, participants take a photo of all meals during the 14 days.

Continuous glucose measurement:

To measure the continuous glucose levels in blood, participants will wear a continuous glucose monitor for 14 days from the day of breaking the fast. To do this, a sensor with a fine filament similar to a needle is attached to the upper arm, which measures glucose during 24 hours. In study participants for whom the continuous measurement of the ketone bodies is also carried out, the continuous glucose measurement is already carried out from the digestive rest day (see next point).

There may be discomfort associated with wearing the sensor and there is a minimal risk of skin irritation or allergic reactions near the sensor site.

Documentation of ketone bodies in urine:

From the digestive rest day until 14 days after breaking the fast, participants will independently determine the ketone body content of the first morning urine with urine test strips every day and document the result in the Buchinger Wilhelmi Amplius app. The color change of the strip indicates the switch from energy production from glucose to energy production from fat reserves.

Collection of stool samples:

Three stool samples are collected, before the start of fasting, as soon as spontaneous bowel movements begin after fasting, and 14 days after fasting. The stool sample after 14 days must be taken independently with the equipment provided and sent by post to the research department of Buchinger Wilhelmi.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Fasting for 5+ days at the Buchinger Wilhelmi clinic in Überlingen or Marbella
* Age: 18-90 years old
* Signed informed consent

Exclusion Criteria:

* Not able to sign the informed consent
* Diagnosed with cachexia, anorexia nervosa, advanced kidney, liver or cerebrovascular insufficiency.
* Chronic manifest psychical and psychiatric diseases
* Participation in another study
* Pregnancy or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Buchinger Wilhelmi clinic in Überlingen
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body weight | From the fasting start until 3 month after fasting
  Changes in body weight in the three-month period after a 5+ day fasting period according to the Buchinger Wilhelmi fasting program

SECONDARY OUTCOMES:
Glycemic regulation | From the fasting start until 3 months after fasting
  Glycemic regulation will be assessed using glycated hemoglobin (HbA1c) measured in venous and/or capillary blood samples at baseline (D-1), 14 days, 1 month, and 3 months after fasting. In addition, continuous glucose monitoring (CGM) will be used during the 14 days following the fasting period.
Change in systemic inflammation | From the fasting start until 3 months after fasting
  To evaluate changes in systemic inflammation, blood samples will be analyzed for levels of C-reactive protein (CRP) at baseline, and again at 14 days, 1 month, and 3 months after the fasting intervention.
Change in systemic inflammation | From the fasting start until 3 months after fasting
  To evaluate changes in systemic inflammation, blood samples will be analyzed for white blood cell (WBC) counts at baseline, and again at 14 days, 1 month, and 3 months after the fasting intervention.
Eating behaviour | During the first 14 days after fasting
  Eating behaviour will be assessed with the MyFoodRepo smartphone app, used during the 14-day period following fasting, where participants photograph their meals. Macronutrient and micronutrient intake is extracted from the image-based food diary using an automated nutrient database.
Eating behaviour | From the fasting start until 3 months after fasting
  Eating behaviour will be assessed with a structured self-report questionnaire completed at baseline, 14 days, 1 month, and 3 months after fasting, assessing dietary patterns.
Resting energy expenditure | From baseline (D-1) to the last day of fasting (Day 5 to Day 25)
  Resting energy expenditure (REE) will be assessed in the morning, under fasted conditions, with participants lying down, using indirect calorimetry. Measurements will be taken at baseline and on the last day of the fasting period (which ranges from 5 to 25 days depending on individual fasting duration).
Wellbeing | From the fasting start until 3 months after fasting
  Subjective wellbeing will be assessed using the WHO-5 Well-Being Index, a validated 5-item questionnaire with a total score ranging from 0 (worst possible wellbeing) to 100 (best possible wellbeing). The questionnaire will be completed at baseline, 14 days, 1 month, and 3 months after fasting.
Wellbeing | From the fasting start until 14 days after fasting
  To assess subjective wellbeing during the fasting period and in the first 14 days post-fasting, participants will provide daily self-reported wellbeing ratings (non-validated), capturing fluctuations in mood, energy, and physical symptoms.
Lifestyle factors | From the fasting start until 3 months after fasting
  Lifestyle behaviour will be assessed using structured self-report questionnaires administered at baseline, 14 days, 1 month, and 3 months after fasting. Topics include:
  Physical activity (type, frequency, and duration) Sleep quality and duration Eating patterns, including eating windows and fasting behaviour Environmental health behaviours (e.g., time in nature, exposure to daylight) General nutrition and hydration practices
Ketone bodies | From the start of fasting until 2 weeks after fasting
  Ketone body levels will be monitored during the fasting period and for 14 days after fasting. Measurements will be performed primarily via urine ketone test strips (acetoacetate), with some participants also performing capillary blood measurements of β-hydroxybutyrate using handheld meters.
Adipose tissue composition | BIA: baseline (Day -1), Day 14, 1 month, and 3 months after fasting Fat biopsies: before fasting (Day -1) and immediately after fasting (last day of fast)
  Whole-body adipose tissue composition will be assessed using bioelectrical impedance analysis (BIA) at baseline, 14 days, 1 month, and 3 months after fasting. In a subset of participants, subcutaneous adipose tissue biopsies will be collected before fasting (baseline) and immediately after fasting (last day of fast; fasting duration varies between 5 and 25 days) to analyze tissue composition and cellular characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Buchinger Wilhelmi Klinik, Überlingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilhelmi de Toledo F, Grundler F, Sirtori CR, Ruscica M. Unravelling the health effects of fasting: a long road from obesity treatment to healthy life span increase and improved cognition. Ann Med. 2020 Aug;52(5):147-161. doi: 10.1080/07853890.2020.1770849. Epub 2020 Jun 10. PMID 32519900
- [Background] Wilhelmi de Toledo F, Grundler F, Goutzourelas N, Tekos F, Vassi E, Mesnage R, Kouretas D. Influence of Long-Term Fasting on Blood Redox Status in Humans. Antioxidants (Basel). 2020 Jun 6;9(6):496. doi: 10.3390/antiox9060496. PMID 32517172
- [Background] Wilhelmi de Toledo F, Grundler F, Bergouignan A, Drinda S, Michalsen A. Safety, health improvement and well-being during a 4 to 21-day fasting period in an observational study including 1422 subjects. PLoS One. 2019 Jan 2;14(1):e0209353. doi: 10.1371/journal.pone.0209353. eCollection 2019. PMID 30601864
- [Background] Scharf E, Zeiler E, Ncube M, Kolbe P, Hwang SY, Goldhamer A, Myers TR. The Effects of Prolonged Water-Only Fasting and Refeeding on Markers of Cardiometabolic Risk. Nutrients. 2022 Mar 11;14(6):1183. doi: 10.3390/nu14061183. PMID 35334843
- [Background] Mesnage R, Grundler F, Schwiertz A, Le Maho Y, Wilhelmi de Toledo F. Changes in human gut microbiota composition are linked to the energy metabolic switch during 10 d of Buchinger fasting. J Nutr Sci. 2019 Nov 12;8:e36. doi: 10.1017/jns.2019.33. eCollection 2019. PMID 31798864
- [Background] Laurens C, Grundler F, Damiot A, Chery I, Le Maho AL, Zahariev A, Le Maho Y, Bergouignan A, Gauquelin-Koch G, Simon C, Blanc S, Wilhelmi de Toledo F. Is muscle and protein loss relevant in long-term fasting in healthy men? A prospective trial on physiological adaptations. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1690-1703. doi: 10.1002/jcsm.12766. Epub 2021 Oct 20. PMID 34668663
- [Background] Muller H, de Toledo FW, Resch KL. Fasting followed by vegetarian diet in patients with rheumatoid arthritis: a systematic review. Scand J Rheumatol. 2001;30(1):1-10. doi: 10.1080/030097401750065256. PMID 11252685
- [Background] Grundler F, Plonne D, Mesnage R, Muller D, Sirtori CR, Ruscica M, Wilhelmi de Toledo F. Long-term fasting improves lipoprotein-associated atherogenic risk in humans. Eur J Nutr. 2021 Oct;60(7):4031-4044. doi: 10.1007/s00394-021-02578-0. Epub 2021 May 7. PMID 33963431
- [Background] Grundler F, Mesnage R, Michalsen A, Wilhelmi de Toledo F. Blood Pressure Changes in 1610 Subjects With and Without Antihypertensive Medication During Long-Term Fasting. J Am Heart Assoc. 2020 Dec;9(23):e018649. doi: 10.1161/JAHA.120.018649. Epub 2020 Nov 23. PMID 33222606
- [Background] Gabriel S, Ncube M, Zeiler E, Thompson N, Karlsen MC, Goldman DM, Glavas Z, Beauchesne A, Scharf E, Goldhamer AC, Myers TR. A Six-Week Follow-Up Study on the Sustained Effects of Prolonged Water-Only Fasting and Refeeding on Markers of Cardiometabolic Risk. Nutrients. 2022 Oct 15;14(20):4313. doi: 10.3390/nu14204313. PMID 36296997
- [Background] Drinda S, Grundler F, Neumann T, Lehmann T, Steckhan N, Michalsen A, Wilhelmi de Toledo F. Effects of Periodic Fasting on Fatty Liver Index-A Prospective Observational Study. Nutrients. 2019 Oct 30;11(11):2601. doi: 10.3390/nu11112601. PMID 31671589
- [Background] Buono R, Longo VD. When Fasting Gets Tough, the Tough Immune Cells Get Going-or Die. Cell. 2019 Aug 22;178(5):1038-1040. doi: 10.1016/j.cell.2019.07.052. PMID 31442398
- [Background] Beck RW, Calhoun P, Kollman C. Use of continuous glucose monitoring as an outcome measure in clinical trials. Diabetes Technol Ther. 2012 Oct;14(10):877-82. doi: 10.1089/dia.2012.0079. PMID 23013201